CLINICAL TRIAL: NCT02308189
Title: Novel Exercise Interventions to Improve Trunk Muscle Function: A Pilot Study
Brief Title: The Back Exercises to Neutralize Disability Study
Acronym: BEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14F025; 1R21AR063909 (NIH)
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Results first posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Low Back Pain
Keywords: Exercise
MeSH Terms: conditions — Low Back Pain; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Active Comparator): Low load resistance exercise training
  Interventions: Behavioral: Exercise
- Exercise with blood flow restriction (Experimental): Low load resistance exercise training with blood flow restriction
  Interventions: Behavioral: Exercise with blood flow restriction

INTERVENTIONS:
Behavioral: Exercise with blood flow restriction — Low load resistance exercise performed with an external pressure cuff applied over both legs or both arms during respective leg and arm exercises.
  Other Names: Kaatsu Training with Blood Flow Restricted Exercise
  Arms: Exercise with blood flow restriction
Behavioral: Exercise — Low load resistance exercise performed with no external pressure cuff applied to the appendicular limbs.
  Other Names: Resistance exercise
  Arms: Exercise

SUMMARY:
A pilot randomized control trial (RCT) to generate effect sizes on the effects of blood flow restricted exercise on trunk extensor cross-sectional area (primary outcome), strength and endurance, whole body and regional lean mass and bone density, as well as the rate of recurrence of LBP (secondary outcomes).

DETAILED DESCRIPTION:
This is a single-blinded, comparison-control group, single-center study of the effects of exercise with and without blood flow restriction applied to the appendicular limbs on safety, body composition (i.e., muscle mass), muscle strength, muscle endurance, whole body and regional lean mass and bone density, and back pain and disability in male and female subjects aged 18-50 years with recurrent low back pain and poor to moderate trunk extensor muscle endurance.

Up to 50 subjects (2 arms) will be randomized in a 1:1 ratio to receive 10-weeks of resistance exercise training with (group 1) or without blood flow restriction (group 2). Randomization will be stratified by sex.

This study will have a screening period of 21 days (day -21 to day -1, screening and baseline measures), a 10-week exercise treatment period (day 1 to day 70) and a 36-week follow up period after the last exercise session (day 70 to day 322). The total duration of the study from first exercise session will be approximately 46 weeks. Baseline measures for muscle size (via MRI), muscle strength, muscle endurance, whole body and regional lean mass and bone density (via DEXA), and measures of back pain and disability will be obtained between day -21 to -1.

Primary Endpoint: The primary endpoint is percent change in trunk extensor muscle cross-sectional area measured by MRI at week 10 (study day 70) after start of exercise training.

Secondary: The secondary endpoints include:

* Muscle strength
* Muscle endurance (time to task failure)
* Whole body and regional lean mass by DEXA
* Whole body and regional bone density by DEXA
* Pain
* Disability
* Safety
* Treatment acceptability Procedures and Assessments Efficacy measures (MRI, muscle strength, muscle endurance, lean mass, bone density, pain, and disability) will be obtained at screening and at week 10 (day 70) and week 20 (day 154).

Safety of blood flow restricted exercise will be assessed based on adverse event findings and monitoring. Subjects will be asked to monitor and report all adverse events (AEs) experienced from the time the informed consent is signed until the end-of-study visit.

Treatment acceptability will be determined by administering the Treatment Evaluation Inventory survey at the end of the fourth and sixteenth exercise sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 50 years, with no significant health issues or conditions that, in the investigator's opinion, would limit the subject's ability to complete the study per protocol or that would impact the capability to get an accurate measurement of study endpoints.
2. Answer yes to the following question: Have you had two or more episodes of low back pain in the past 12-months with at least one of the episodes causing a restriction of work or leisure time activity?
3. Exhibit low trunk extensor endurance defined as the time to task failure during the modified-Sorenson test of less than 176 seconds.
4. Body mass index (BMI) between 19 and 37 kg/m2 inclusive.
5. With no condition that could limit participation in supervised resistance training exercise based on the Physical Activity Readiness Questionnaire (PAR-Q) (i.e., if a study participant answers yes to questions 1-4 they will be excluded, if they answer yes to 5-7 they will require clearance for participation by the study physician).
6. Sedentary lifestyle defined by a classification of "low" or "moderate" levels of physical activity based on the scoring criteria for the International Physical Activity Questionnaire (IPAQ).
7. Willing to maintain current diet and adhere to exercise programs described for the study and to not start any new dieting/weight management programs.
8. Willing and able to return for all clinic visits and complete all study-related procedures.
9. Able to read, understand, and complete study-related questionnaires
10. Able to read and understand, and willing to sign the informed consent form (ICF).

Exclusion Criteria:

1. Participation in progressive resistance exercise within the previous 24 weeks prior to screening.
2. Participation in any clinical trial within 24 weeks prior to screening.
3. Hospitalization (medical confinement for ≥24 hours), or immobilization, or major surgical procedure requiring general anesthesia within 24 weeks prior to screening, or any planned surgical procedures during the study period.
4. Limb amputation (except for toes) and/or any fracture within 24 weeks.
5. Osteoarthritis, rheumatologic diseases or orthopedic disorders which will not allow completion of the motions required for the resistance exercise.
6. Conditions (such as myasthenia gravis, myositis, muscular dystrophy or myopathy, including drug-induced myopathy) leading to muscle loss, muscle weakness, muscle cramps or myalgia.
7. Chronic or relapsing/remitting gastrointestinal disorders such as inflammatory bowel diseases, irritable bowel syndrome or gastrointestinal infections within 28 days of screening.
8. Acute viral or bacterial upper or lower respiratory infection at screening
9. Moderate or severe chronic obstructive pulmonary disease.
10. Back pain greater than 4 (on a 10 point numeric pain rating scale) at screening
11. Leg length discrepancy > 3 cm.
12. Current or recent (i.e., within 12 weeks) of narcotics or muscle relaxants.
13. Currently pregnant (confirmed via a urine test) or planning to become pregnant within the next year at screening.
14. Report unexplained weight loss over the past 30 days (> 10 pounds).
15. Report having pending litigation related to low back pain or currently receiving disability for low back pain.
16. Report having received treatment for low back pain from a health care practitioner in the past 6 weeks.
17. History of spine surgery or hip arthroplasty.
18. Cancer requiring treatment currently or in the past 3 years (except primary non-melanoma skin cancer or in situ cervical cancer)
19. Moderate or severe asthma with current or recurring symptoms within the last 1-year.
20. Known history of human immunodeficiency virus (HIV) antibody and/or positive hepatitis B surface antigen (HBsAg) and/or positive hepatitis C antibody (HCV) at screening.
21. Neurological conditions resulting in impaired muscle function or mobility (e.g., stroke with residual paresis, paralysis, multiple sclerosis, or Parkinson Disease).
22. Psychiatric conditions that warrant acute or chronic therapeutic intervention (e.g., major depressive disorder, bipolar disorder, panic disorder, schizophrenia) that in the investigators opinion may interfere with the conduct of study procedures
23. History of cardiac conditions such as heart failure (NYHA class II-IV), angina (including unstable angina), myocardial infarction, cardiomyopathy, any cardiac arrhythmia (except stable sinus dysrhythmia or atrial fibrillation) or valvular heart disease (except asymptomatic mitral valve prolapse).
24. History of peripheral vascular disease.
25. Subjects with the following abnormal ECG findings at screening will be excluded:

    Electrocardiogram findings indicative of left ventricular hypertrophy (LVH) (based on Cornell voltage criteria): For men: S in V3 plus R in a VL >2.8 mV (28 mm) For women: S in V3 plus R in a VL >2.0 mV (20 mm) Electrocardiogram finding of QT prolongation defined as QTcF > 470 ms
26. Diabetics using insulin are excluded.
27. Abnormal or uncontrolled blood pressure at the screening visit defined as diastolic BP >100 and/or systolic BP >160 mm Hg; if taking anti-hypertensive medication, have to be on stable doses of medication for more than 3 months.
28. Current or recent history (within 1 year of screen) of heavy alcohol consumption (males ≥ 21 drinks/week, 4 drinks/day; females ≥ 14 drinks/week, 3 drinks/day) or drug abuse.
29. Current or previous use of any drugs known to influence muscle mass or performance within 24 weeks. These may include, but are not limited to, anabolic steroids, IGF-1, growth hormone (GH), replacement androgen therapy, anti-androgen therapy.
30. Use of systemic glucocorticoids within 12 weeks prior to screening.
31. Having body dimensions that exceed the MRI or exercise equipment limits.
32. Unable to undergo MRI (e. g. body containing any metallic medical devices or equipment, including heart pacemakers, metal prostheses, implants or surgical clips, any prior injury from shrapnel or grinding metal, exposure to metallic dusts, metallic shavings or having tattoos containing metallic dyes).
33. Unable to reliably undergo exercise or strength tests described for this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-12; Primary Completion 2016-11-24 (Actual); Study Completion 2017-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Clark, PhD, Principal Investigator — Ohio Musculoskeletal and Neurological Institute (OMNI)
Locations (1):
- Ohio Musculoskeletal and Neurological Institute (OMNI) at Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amano S, Ludin AF, Clift R, Nakazawa M, Law TD, Rush LJ, Manini TM, Thomas JS, Russ DW, Clark BC. Effectiveness of blood flow restricted exercise compared with standard exercise in patients with recurrent low back pain: study protocol for a randomized controlled trial. Trials. 2016 Feb 12;17:81. doi: 10.1186/s13063-016-1214-7. PMID 26867541

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise | Exercise With Blood Flow Restriction
Started | 17 | 15
Completed | 16 | 14
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: a total of 32 participants were randomized, 2 were withdrawn after randomization
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise | Exercise With Blood Flow Restriction | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Categorical [Count of Participants; unit: Participants] — Population: Two subjects withdrew after randomization. Analysis completed on 30 subjects
  Participants
    number analyzed (Participants) | 16 | 14 | 30
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 16 | 14 | 30
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (10.3) | 28.4 (9.2) | 29.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 7 | 5 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Trunk Extensor Muscle Cross Sectional Area % of Change
Description: The primary endpoint is percent change in trunk extensor muscle cross-sectional area measured by The primary endpoint is percent change in trunk extensor muscle cross-sectional area measured by MRI at week 10 (study day 70) after start of exercise training.
Time Frame: Baseline and following 10-weeks of exercise training. Values are calculated from % change.
Population: Per protocol analysis of completed study participants
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Exercise | Exercise With Blood Flow Restriction
Number analyzed (Participants) | 16 | 14
percentage of change | -1.7 (1.0) | -3.9 (0.9)

2. Secondary Outcome: Muscle Strength % of Change
Description: Maximal muscle strength
Time Frame: Baseline and following 10-weeks of exercise training. Values calculated are % of change
Population: Study participants completing study.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Exercise | Exercise With Blood Flow Restriction
Number analyzed (Participants) | 16 | 14
percentage of change from baseline | 8.4 (3.1) | 4.7 (2.2)

3. Secondary Outcome: Muscle Endurance (Time to Task Failure) % of Change
Description: Time for successfully performing a sustained, submaximal muscle contraction
Time Frame: Baseline and following 10-weeks of exercise training. Values are calculated on % of change.
Population: Study participants completing study.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Exercise | Exercise With Blood Flow Restriction
Number analyzed (Participants) | 16 | 14
percentage of change from baseline | 25.1 (4.9) | 21.0 (5.1)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and assessed for each subject for 9-months
Description: AE definitions followed clinicaltrials.gov definitions.
Arm/Group | Exercise | Exercise With Blood Flow Restriction
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 0/17 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes